CLINICAL TRIAL: NCT05827588
Title: A Prospective, Single-arm Study to Evaluate the Feasibility of Automated Wearable Artificial Kidney Peritoneal Dialysis (AWAK PD) in Subjects With End-Stage Kidney Disease
Brief Title: Late Feasibility Study to Evaluate Safety and Efficacy of AWAK PD Device in Subjects With ESKD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AWAK Technologies Pte Ltd (Industry)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG-CLI-DOC-445
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Peritoneal dialysis; Wearable medical device; Home-based therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AWAK PD (Experimental): Wearable/Ultra-portable peritoneal dialysis device for home-use
  Interventions: Device: AWAK PD

INTERVENTIONS:
Device: AWAK PD — Daily 7- or 9-hour therapy (with or without a last fill) that is a form of automated peritoneal dialysis being done by subjects who are already on daily PD therapy

SUMMARY:
The goal of this late feasibility clinical trial is to evaluate the safety and effectiveness of the Automated Wearable Artificial Kidney (AWAK) peritoneal dialysis (PD) device in subjects with end-stage kidney disease. The main questions it aims to answer are:

* the success of AWAK PD therapies when used in a home-setting
* the safety and effectiveness of the AWAK PD system

Participants will:

* be titrated to find a suitable AWAK PD prescription
* be trained on how to use the AWAK PD system independently
* use the AWAK PD system at home for at least 7 days

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study.
2. Male or female ≥22 years of age.
3. Treated with PD for at least 3 months before Screening.
4. Has weekly Kt/Vurea (renal + peritoneal) ≥1.7
5. No acute peritonitis, catheter infection, exit site, or subcutaneous tunnel infection within 3 months before Screening.

Exclusion Criteria:

1. Severe comorbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the subject to be a good investigation candidate
2. Recent (within the previous 6 months) history of major cardiovascular events (e.g., stroke, acute myocardial infarction).
3. Diagnosed with New York Heart Association (NYHA) Class III or Class IV heart failure.
4. Poorly controlled diabetes mellitus as defined by hemoglobin A1c >9.0% during Screening
5. Subject has a current abdominal hernia.
6. Subject has an active infection requiring systemic antibiotics or antifungal therapy.
7. Active infection of hepatitis B and C, or HIV infection at any time.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Proportion of completed therapies | 7 days

SECONDARY OUTCOMES:
Proportion of subjects maintaining body weight within ±5% of the subject's target weight | 7 days
Change in serum levels of markers of uremia (urea and creatinine) | 7 days
Proportion of subjects maintaining serum sodium and potassium levels within normal clinical ranges | 7 days
Incidence of serious adverse events (SAEs), serious adverse device effects (SADEs), adverse events (AEs), adverse device effects (ADEs), and device deficiency events | 7 days
Incidence of peritonitis related to the use of AWAK PD | 30 days
Change in the incidence and severity of dialysis-related signs and symptoms based on responses on the PD Dialysis Symptoms Questionnaire | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Foo, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No